CLINICAL TRIAL: NCT03675204
Title: Establishment of the Breast Milk Database in China
Status: Completed | Type: Observational
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-SC-05-FC-001
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2018-09

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — A minimum of 60ml of breast milk will be collected for each subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Collect breast milk samples in various administrative regions of China to measure the nutrients in breast milk; analyze the composition of nutrients; and establish the database of breast milk in China.

DETAILED DESCRIPTION:
The study cities are Guangzhou, Weihai, Chengdu, Beijing, Harbin, Wuhan, Jinhua, Zhengzhou and Lanzhou.

Breast milk will be collected at 9:00-11:00 in the morning from 15 to180 days after giving birth. The nutrients (protein, triglyceride, phospholipid, oligosaccharides and probiotics) in the collected breast milk samples will be measured. These data will be used to establish the breast milk database in China. This databased will provide references for infant nutrient intake and for the formulation and revision of infant formula standards. It will also provide references for the development of new infant formula products in China.

ELIGIBILITY:
Inclusion Criteria:

* Lactating mother 25 ~ 35 years old;
* Breast-feeding infants (15 ~180 days old );
* Physically healthy by self-evaluation;
* Does not smoke;
* Does not drink alcohol;
* Have given birth to physically healthy infants;
* Signed the informed consent forms.

Exclusion Criteria:

* Being treated for gastrointestinal symptoms;
* Suffering from mastitis;
* Suffering from infectious diseases (tuberculosis, viral hepatitis and HIV infection);
* Suffering from cardiovascular disease;
* Suffering from metabolic diseases (such as diabetes);
* Suffering from mental system diseases;
* Suffering from cancer and other malignant diseases;
* Having history of taking antibiotics;
* Not able to answer the study questions;
* Participating in any nutritional or pharmaceutical intervention study recently.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy lactating mother of 25 ~ 35 years old who are currently breast-feeding infants of 15 ~180 days old. Subjects are equally distributed in the postpartum time period of 15~35 days, 36~65 days, 66~95 days, 96~125 days, 126~55 days and 156~185 days
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Protein in breast milk | At enrollment
  Protein in breast milk measured in percent (%)

SECONDARY OUTCOMES:
Osmotic pressure | At enrollment
  Osmotic pressure (mmolOsm/Lkg.H2O) in breast milk
Fatty acids in breast milk | At enrollment
  Fatty acids composition (mg/L) in breast milk
Amino acids | At enrollment
  Amino acids composition (mg/L) in breast milk
Oligosaccharides | At enrollment
  Oligosaccharides levels (mg/L) in breast milk
Probiotics | At enrollment
  Probiotics composition (species) measured using gene sequencing in breast milk;
Vitamins | At enrollment
  Vitamins composition (μg/L) in breast milk
Minerals | At enrollment
  Minerals composition (mg/L) in breast milk
Hormones | At enrollment
  Hormones composition (mg/L) in breast milk
Dietary composition of participating mothers | At enrollment
  Investigation on the dietary composition of participating mothers obtained using questionnaire
Height of participating mothers | At enrollment
  Height measurement (cm) of participating mothers
Weight of participating mothers | At enrollment
  Body weight measurement (kg) of participating mothers
Age of participating mothers | At enrollment
  Age (years) of participating mothers obtained using questionnaire
Educational level of participating mothers | At enrollment
  Educational level of participating mothers obtained using questionnaire
Occupation of participating mothers | At enrollment
  Occupation of participating mothers obtained using questionnaire
Physical health condition of participating mothers | At enrollment
  Physical health condition of participating mothers assessed by questionnaire
Triglyceride | At enrollment
  Triglyceride (mg/g) contents in breast milk
Phospholipid | At enrollment
  Phospholipid (mg/g) contents in breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Shilong Jiang, Study Director — Heilongjiang Feihe Dairy Co. Ltd.